CLINICAL TRIAL: NCT07310992
Title: The Effect of Meditation Practice Combined With Cardiac Rehabilitation on Improving Quality of Life and Controlling Blood Pressure.
Brief Title: Effect of Meditation as an Adjunct to Cardiac Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Guacira Grecca, Guacira Grecca, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91829725.6.0000.5462
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: High Blood Pressure (& [Essential Hypertension]); Meditation Training; Rehabilitation Exercise
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Arm 1 - Control Group
  Name: Standard Cardiac Rehabilitation
  Description:
  Participants undergo 60 minutes of aerobic and resistance training, twice per week, for 12 weeks, with optimized medical therapy.
  Intervention Type: Behavioral / Exercise Duration: 12 weeks
  Arm 2 - Meditation Group (Intervention Group)
  Name: Cardiac Rehabilitation + Meditation
  Description:
  Participants undergo 60 minutes of aerobic and resistance training + 15 minutes of guided mindfulness meditation at the end of each session, twice per week, for 12 weeks, with optimized medical therapy.
  Intervention Type: Behavioral / Meditation (Mindfulness) Duration: 12 weeks
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Meditation + Rehabilitation (Experimental): Participants in this group will undergo the standard cardiac rehabilitation program consisting of 60 minutes of aerobic and resistance training, twice a week for 12 weeks. Additionally, they will participate in a 15-minute voice-guided mindfulness meditation session immediately following each exercise session. Participants also receive optimized medical therapy.
  Interventions: Behavioral: Meditation
- Active Comparator: Standard Rehabilitation (Active Comparator): Participants in this group will undergo the standard cardiac rehabilitation program consisting of 60 minutes of aerobic and resistance training, twice a week for 12 weeks, along with optimized medical therapy. This group does not receive the guided meditation intervention.
  Interventions: Procedure: Standard Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Meditation — Participants in this group will undergo the standard cardiac rehabilitation program consisting of 60 minutes of aerobic and resistance training, twice a week for 12 weeks. Additionally, they will participate in a 15-minute voice-guided mindfulness meditation session immediately following each exercise session. Participants also receive optimized medical therapy.
  Arms: Experimental: Meditation + Rehabilitation
Procedure: Standard Cardiac Rehabilitation — Participants in this group will undergo the standard cardiac rehabilitation program consisting of 60 minutes of aerobic and resistance training, twice a week for 12 weeks, along with optimized medical therapy. This group does not receive the guided meditation intervention.
  Arms: Active Comparator: Standard Rehabilitation

SUMMARY:
Cardiovascular rehabilitation is a well-established standard of care that significantly reduces morbidity and mortality while improving quality of life. However, integrating behavioral interventions into physical training may offer additional benefits for autonomic regulation and emotional well-being.

This randomized clinical trial aims to investigate the efficacy of adding a brief, guided mindfulness meditation session to a standard cardiovascular rehabilitation program. The study seeks to determine whether this combined intervention enhances blood pressure control, improves perceived quality of life, and increases patient adherence compared to standard rehabilitation alone.

Participants newly enrolled in the Cardiac Rehabilitation Service will be randomized into two groups. Both groups will undergo a standard 12-week regimen of aerobic and resistance training combined with optimized medical therapy. The intervention group will additionally receive 15 minutes of voice-guided mindfulness meditation at the end of each exercise session. Key outcome measures include blood pressure variability, quality of life scores (assessed via EQ-5D), and attendance rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 years or older.
* Newly enrolled in the Phase II Cardiac Rehabilitation Program.
* Clinically stable condition with medical clearance to perform aerobic and resistance exercises.
* Diagnosis of cardiovascular disease (e.g., coronary artery disease, post-myocardial infarction, post-cardiac surgery, or stable heart failure) warranting rehabilitation.
* Willingness and cognitive ability to provide written informed consent.
* Availability to attend the twice-weekly sessions for the 12-week duration of the study.

Exclusion Criteria:

* Current regular practice of meditation, yoga, or other mind-body techniques (defined as formal practice more than once a week in the previous 3 months).
* Current participation in other psychological or behavioral intervention clinical trials.
* Severe cognitive impairment or psychiatric disorders that preclude understanding of the meditation instructions or group participation (e.g., dementia, untreated psychosis).
* Unstable clinical conditions such as unstable angina, uncontrolled arrhythmias, or decompensated heart failure that contraindicate physical exercise.
* Significant orthopedic or neurological limitations that prevent the performance of the exercise protocol.
* Refusal to participate in the randomization process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scores (EuroQol EQ-5D Visual Analogue Scale) | Baseline and Week 12
  Quality of life is assessed using the EuroQol Five Dimensions Questionnaire (EQ-5D). This instrument includes the EQ Visual Analogue Scale (EQ-VAS), a quantitative measure of the participant's self-rated health status. The EQ-VAS scores range from a minimum of 0 to a maximum of 100, where 0 represents 'the worst health you can imagine' and 100 represents 'the best health you can imagine'. Higher scores indicate better health outcomes and higher quality of life.

SECONDARY OUTCOMES:
Change in Systolic and Diastolic Blood Pressure | Baseline and Week 12
  Assessment of both systolic and diastolic blood pressure parameters using a validated digital oscillometric device. Measurements are recorded in millimeters of mercury (mmHg). Reductions in both systolic and diastolic values indicate clinical improvement.
Rate of Rehabilitation Adherence | Through study completion, an average of 12 weeks